CLINICAL TRIAL: NCT00223470
Title: Cytokine Regulation of Periradicular Pain in Humans
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 012-1904-455; K23DE014864-01A1S1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Apical Periodontitis of Pulpal Origin
Keywords: pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sterile paper points are placed in the canal for 30 seconds
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical trial evaluates the role of cytokines in patients needing root canal treatment with diagnosis of necrotic pulp and chronic apical periodontitis

DETAILED DESCRIPTION:
This study evaluates whether periradicular exudate concentrations of cytokines differ in patients experiencing pain and mechanical allodynia due to pulpal necrosis with an acute exacerbation of a chronic apical periodontitis, as compared to patients with pulpal necrosis with chronic apical periodontitis, but no pain or mechanical allodynia

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 16 years of age.
2. Clinical indication for Non-Surgical Root Canal Therapy (NSRCT).
3. 1st or 2nd maxillary or mandibular molar
4. Diagnosis must be Chronic Apical Periodontitis (CAP) with or without symptoms.
5. Intact, mature apices.
6. ASA I or II

Exclusion Criteria:

1. Failure to meet any of the above
2. Previous NSRCT
3. Previous pulpotomy or pulpectomy
4. Suppurative apical periodontitis
5. Patients taking medications which can affect their pain rating or medications which effect their immune system ( such as glucocorticoids)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to the Endodontics department with an indication for root canal treatment
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asma A Khan, BDS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Univerity of Texas Health Science Center at San Antonio, San Antonio, Texas, United States